CLINICAL TRIAL: NCT01217216
Title: Cancer Survival Through Weight Loss and Exercise (CASTLE)
Brief Title: Cancer Survival Through Weight Loss and Exercise
Acronym: CASTLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 28036
Record Dates: First submitted 2010-10-05; First posted 2010-10-08 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Survivors
Keywords: Breast Cancer; Weight loss; Group Intervention; Telephone Intervention
MeSH Terms: conditions — Breast Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group-based Intervention (Active Comparator): We randomly assigned 30 individuals to a group-based intervention to promote weight loss through dietary restriction and physical activity.
  Interventions: Behavioral: Group-based Intervention
- Telephone-based Intervention (Active Comparator): We randomly assigned 22 individuals to the telephone-based intervention to promote weight loss through dietary restriction and physical activity.
  Interventions: Behavioral: Telephone-based Intervention

INTERVENTIONS:
Behavioral: Group-based Intervention — compared effects of a group-based intervention on weight loss and physical activity.
  Arms: Group-based Intervention
Behavioral: Telephone-based Intervention — compared telephone-based intervention to weight loss and physical activity.
  Arms: Telephone-based Intervention

SUMMARY:
To test the effectiveness and feasibility of intensive motivational, behavior modifying intervention aimed at improving physical activity and dietary habits to produce at least 7% weight loss in women with a history of breast cancer in a community health setting.

DETAILED DESCRIPTION:
This study will be divided into two phases (Phase I and II) that will differ by the intensity of motivational intervention. In Phase I, participants will receive 6 months of intensive weekly group-based or telephone-based motivational, behavior modifying intervention aimed at improving physical activity levels and dietary habits. Phase II will be an additional 6 months of monthly individualized motivational intervention in order to attain and maintain at least 7% body weight loss. All participants will attend an orientation, 2 run-in sessions, and a baseline assessment prior to the intervention. Participants will then be assigned to either the group based intervention or telephone intervention. The first 30 participants will enter into the group-based intervention and the second 30 will enter into the telephone-based intervention. Follow-up visits will be completed at the end of Phase I (week 25) and Phase II (week 50). Up to 60 women with a previous history of breast cancer will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 30 and 75.
* Positive history of breast cancer treatment completed at least 2 months but no longer than 36 months prior to randomization.
* BMI ≥ 25 kg/m2 and ≤ 45 kg/m2
* Not involved in regular physical activity or weight loss management programs.
* Stage I, II or IIIa breast cancer with good prognosis.

Exclusion Criteria:

* Presence of any co-morbidities including cardiovascular disease or diabetes
* Fasting triglycerides > 500 mg/dl.
* Consume more than 14 alcoholic beverages per week.
* A history of drug abuse, or excess alcohol consumption (40g/day)6.
* Currently dieting or engaging in any activity with the goal of losing weight.
* Significant intentional weight loss in the past year (> 50 lbs in the past year) or current use of weight loss medications.
* History of gastrointestinal bypass or other bariatric surgery in the last 3 years.
* Pregnant or plan on becoming pregnant in the next 12 months.
* Factors that may limit adherence to intervention or affect conduct of the trial.
* Unable or unwilling to communicate with staff, to provide written informed consent, or accept the randomized assignment.
* Failure to complete run-in and baseline testing.
* Lack support from health care provider or family members.
* Other temporary intervening event, such as sick spouse, bereavement, or recent move.
* Any other medical condition or disease that is life threatening or that can interfere with or be aggravated by exercise.
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder.
* Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 year
  To examine the effectiveness of using motivational, behavioral interventions aimed at improving physical activity levels and dietary habits to produce weight loss in women with a history of breast cancer.

SECONDARY OUTCOMES:
Feasibility of recruiting breast cancer survivors | 1 year
  To examine the feasibility of recruiting, administering, and maintaining interventions in a small sample of women with a history of breast cancer in a community health setting for pilot data.
Examination of health outcomes, breast cancer reoccurrence, and mortality. | 1 year
  To examine health outcomes, cancer reoccurrence, and mortality in women with a history of breast cancer within the 12 month period via adverse events. Additional procedures include resting ECG, waist circumference, weight, and blood work.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Church, MD, MPH, PhD, Principal Investigator — Pennington Biomedica Research Center; Donna H Ryan, MD, Study Director — Pennington Biomedical Research Center; Conrad P Earnest, PhD, Study Director — Pennington Biomedical Research Center; Valerie H Myers, PhD, Study Director — Pennington Biomedical Research Center; Catherine M Champagne, PhD, Study Director — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Harris MN, Swift DL, Myers VH, Earnest CP, Johannsen NM, Champagne CM, Parker BD, Levy E, Cash KC, Church TS. Cancer survival through lifestyle change (CASTLE): a pilot study of weight loss. Int J Behav Med. 2013 Sep;20(3):403-12. doi: 10.1007/s12529-012-9234-5. PMID 22535636